CLINICAL TRIAL: NCT03647098
Title: Survival Outcomes for Lung Cancer
Brief Title: Survival Outcomes of Lung Cancer
Acronym: Soul
Status: Recruiting | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Director of Clinical Trial Center, Hunan Province Tumor Hospital
Other Study IDs: 20180176
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue were obtained with the permission from patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Cohorts 1: Non-small cell lung cancer patients with EGFR mutations. Group A ： Single EGFR Drive gene Mutations Group B ：EGFR co-mutant with De novo MET alterations Group C ：EGFR co-mutant with other genes including ALK , ROS , RET , BRAF .etc
  Interventions: Drug: Treatment
- Cohorts 2: Non-small cell lung cancer patients with ALK-fusion positive.
  Interventions: Drug: Treatment
- Cohorts 3: Non-small cell lung cancer patients with ROS-1-positive.
  Interventions: Drug: Treatment
- Cohorts 4: Non-small cell lung cancer patients with Other Rare Mutations.
  Interventions: Drug: Treatment
- Cohorts 5: Driver-negative lung cancer patients with ADC and SQC.
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment — Treatment decisions guided by molecular profiling and clinical judgment of principal investigators

SUMMARY:
This is a prospective study to analyze the survival outcomes of different groups about lung cancer patients.

DETAILED DESCRIPTION:
This study aims to analyze the survival outcomes of different groups about lung cancer patients. All the groups were assessed to the treatment decisions guided by molecular profiling and clinical judgment of principal investigators

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements and contents of the clinical trial .
2. Age ≥ 18 years.
3. Histopathology or cytology confirmed lung cancer
4. ECOG <=2.
5. Predicted survival ≥ 12 weeks.
6. Adequate bone marrow hematopoiesis and organ function
7. Presence of measurable lesions according to RECIST 1.1.

Exclusion Criteria:

1. Subjects who have received any of the following treatments must be excluded:

   * Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
   * Ongoing (or inability to discontinue) possibly potent CYP1A2, CYP3A inhibitor (1 week), or inducer (2 weeks) drug therapy or herbal supplements within 1-2 weeks prior to the first dose.
2. Presence of spinal cord compression or meningeal metastasis.
3. History of other malignant tumors within 2 years.
4. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
5. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
6. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
7. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
8. Heart-related diseases or abnormalities
9. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
10. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb drugs due to previous bowel resection.
11. Live vaccine was given 2 weeks before the first medication.
12. Women who are breastfeeding or pregnant.
13. Hypersensitivity to the test drug and the ingredients.
14. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung cancer
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 5 years
  PFS defines as first dose to first documented disease progression assessed by investigator or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Time from first subject dose to study completion, or up to 5 years
  To assess overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)
Adverse events (AEs) | Time from first subject dose to study completion, or up to 5 years
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — zhangyongchang@csu.edu.cn
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No